CLINICAL TRIAL: NCT00838409
Title: Examination of Metabolic Determinants of Behavior and Motivation in Obesity: Implication to the Development of New Strategies for Achieving Body Weight Health
Brief Title: USDA Behavior, Motivation & Nutrition Study
Status: Completed | Type: Observational
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: WHNRC003
Record Dates: First submitted 2009-02-04; First posted 2009-02-06 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Body Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and saliva samples will be kept for future research purposes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This study will be a cross-sectional study. The primary aim of this study is to compare the relationship between neurological function, metabolic measures and health-related behaviors between normal weight and overweight/obese perimenopausal women.

DETAILED DESCRIPTION:
To examine physiological and behavioral factors that may help determine health in perimenopausal middle age women. Neuroendocrine function will be measured by broad assessment of hypothalamic-pituitary-adrenal (HPA) activity. We will also assess metabolic profiles and behavioral and emotional function. We plan to determine correlations between these measures and nutritional state. Other measures may include insulin, glucose, leptin, IGF-1, triglycerides, free fatty acids, and ghrelin and eating attitudes and physical reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass index 18-39.9 kg/m2
* Peri-menopausal status by self-report

Exclusion Criteria:

* Pregnant
* Plan to become pregnant
* Breastfeeding in the last 6 months
* Multiple sclerosis, amyotrophic lateral sclerosis, Parkinson's disease
* Menopause confirmed
* Unable to refrain from smoking for five hours (self-report)
* Unable to refrain from consuming alcohol for two days (self-report)
* Weight change > 10 lbs in the preceding 6 months
* Chronic corticosteroid use
* Oral corticosteroids used more than twice in the last 12 months
* Hormonal contraceptives
* Antipsychotic, anti-anxiety and anti-depressant medications
* Beta adrenergic blockers
* Sibutramine, orlistat, phentermine, phendimetrazine, topiramate, zonisamide
* Immunosuppressants
* Amphetamines and other stimulants
* Severe food allergies or intolerances to foods
* Insulin Dependent Diabetes Mellitus

Ages: 42 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Correlation between metabolic measures and health-related behaviors in normal weight and overweight/obese perimenopausal women. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Laugero, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- See also: USDA, ARS, WHNRC — http://www.ars.usda.gov/main/site_main.htm?modecode=53062500